CLINICAL TRIAL: NCT03852589
Title: Comparison of C-MAC Videolaryngoscopy-guided Proseal Laryngeal Mask Airway Placement vs Conventional Blind Technique: a Prospective Randomized Study
Brief Title: The Effect of Placement of Proseal Laryngeal Mask Airway With C-Mac Videolaryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ülkü Özgül, Associate professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: UlkuVL
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Laryngeal Masks; Anesthesia, General; Videolaryngoscopy
Keywords: Airway management; Videolaryngoscopy; General anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-MAC Videolaryngoscope (Active Comparator): C-MAC Videolaryngoscope: An intubating device that is used for endotracheal intubation. Proseal laryngeal mask airway will be inserted with C-MAC Videolaryngoscope
  Interventions: Device: C-MAC videolaryngoscope
- Blind (Active Comparator): Proseal laryngeal mask airway will be inserted with digital finger
  Interventions: Device: Blind

INTERVENTIONS:
Device: C-MAC videolaryngoscope — An intubating device that is used for endotracheal intubation. PLMA will inserted by anesthesiologist with C-MAC videolaryngoscope.
  Arms: C-MAC Videolaryngoscope
Device: Blind — PLMA will inserted by anesthesiologist with digital finger.
  Arms: Blind

SUMMARY:
The ProSeal laryngeal mask airway (ProSeal LMA; Intavent Orthofix, Maidenhead, UK) is a device with a double cuff to improve the seal and a drain tube to help prevent aspiration and gastric insufflation, facilitate passage of a gastric tube, and provide information about malposition. The manufacturer recommends inserting the ProSealTM LMA using digital manipulation or with an introducer tool, but both these techniques have lower success rates than the classic LMA.

This prospective study that will investigated the usefulness of the C-MAC videolaryngoscopy for inserting a PLMA in anesthetized non-paralyzed patients and compared it with the index finger.

DETAILED DESCRIPTION:
Airway management is one of the cornerstones for modern anaesthesia and is vital for all patients undergoing general anaesthesia. Supraglottic airway devices (SADs) are increasingly used for managing airways.

The ProSeal laryngeal mask airway (PLMA) (Laryngeal Mask Company, San Diego, CA, USA) is a supraglottic airway device with a larger cuff than the Classic laryngeal mask airway to produce a better seal. The PLMA is also equipped with a drainage tube to permit insertion of a gastric tube and evacuation of gastric content. The presence of the drainage tube reduces the risk of aspiration, which is the major concern of the Classic laryngeal mask airway, especially when the device is used with positive pressure ventilation. While a dedicated introducer (commonly known as an ''introducer tool'') is recommended by the manufacturer to facilitate insertion of the PLMA, difficulties can still be encountered during insertion. The PLMA insertion success rate at first attempt has been reported as 82-87%, which is lower than the insertion success rate of the Classic laryngeal mask airway.

Malpositioning of the PLMA is common in clinical practice because its soft cuff can fold over onto itself. Malpositioning of the device can result in severe leaks and even obstruction of the airway, with potentially negative outcomes for the patient. Although the incidence of complications(e.g. airway trauma, obstruction, regurgitation, gastric distension with mechanical ventilation) is likely to be higher with an incorrectly placed SAD, clinical airway obstruction can result from other causes, such as laryngospasm and transient closure of the glottis.

Many methods have been proposed to facilitate insertion of PLMAs, including insertion of a gastric tube,a suction catheter, or a gum elastic bougie into the drainage tube. These techniques help to prevent the PLMA soft cuff from folding over and help to decrease the incidence of malpositioning.

This prospective study that will investigated the usefulness of the C-MAC videolaryngoscopy for inserting a PLMA in anesthetized non-paralyzed patients and compared it with the index finger.

ELIGIBILITY:
Inclusion Criteria:

* 18- 65 years
* Undergoing short surgical prcedures with general anesthesia using a PLMA
* American Society of Anesthesiology score I-II

Exclusion Criteria:

* Anticipated difficult airway
* Risk of aspiration
* Patients who refused written informed consent forms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
First attempt success rate | From inserted PLMA to seeing meaningful end-tidal carbon dioxide levels up to 2 minutes
  The PLMA will inserted into hypopharynx, the cuff will inflated with an appropraite volume of air. An effective airway will judged by a square wave on capnography.

SECONDARY OUTCOMES:
Insertion time | From inserted PLMA to seeing two meaningful end-tidal carbon dioxide levels up to 3 minutes
  Insertion time was the time between picking up the PLMA and successful placement
Adverse Events | During the first 24 hour postoperatively
  Blood on the surface of the cuff, laryngospasm, hypoxia, hoarseness,sore throat
Fiberoptic Score | After the PLMA insertion up to 5 minutes
  Fiberoptic view of PLMA placement through the airway tube was graded on a scale from 4 (best view) to 1 (worst view)
Airway Sealing Pressure | After the PLMA insertion up to 5 minutes
  Fresh gas flow was adjusted to 3 L/min, and after closing the expiratory valve, the airway pressure at which an audible leak in the mouth was heard will recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ulku Ozgul, Principal Investigator — Inonu University Faculty of Medicine
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koay CK, Yoong CS, Kok P. A randomized trial comparing two laryngeal mask airway insertion techniques. Anaesth Intensive Care. 2001 Dec;29(6):613-5. doi: 10.1177/0310057X0102900609. PMID 11771605
- [Background] Sorbello M, Petrini F. Supraglottic Airway Devices: the Search for the Best Insertion Technique or the Time to Change Our Point of View? Turk J Anaesthesiol Reanim. 2017 Apr;45(2):76-82. doi: 10.5152/TJAR.2017.67764. Epub 2017 Apr 1. PMID 28439437
- [Derived] Ozgul U, Erdil FA, Erdogan MA, Begec Z, Colak C, Yucel A, Durmus M. Comparison of videolaryngoscope-guided versus standard digital insertion techniques of the ProSeal laryngeal mask airway: a prospective randomized study. BMC Anesthesiol. 2019 Dec 30;19(1):244. doi: 10.1186/s12871-019-0915-3. PMID 31888511